CLINICAL TRIAL: NCT01267071
Title: A Single Dose, Open Label, Nonrandomized, Study to Evaluate the Pharmacokinetics and Absolute Bioavailability of GSK962040 Given as an Oral Dose Simultaneously With an Intravenous Microtracer Dose of [14C]-GSK962040 in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Absolute Bioavailability of GSK962040 Given as an Oral Dose Simultaneously With an Intravenous Microtracer Dose of [14C]-GSK962040 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114136
Record Dates: First submitted 2010-11-18; First posted 2010-12-24 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Gastroparesis
Keywords: Entero-test; Phase I; GSK962040; i.v. microtracer; radioactivity; pharmacokinetics; healthy volunteer
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): GSK962040 (50 mg, SD, oral)
  Interventions: Drug: A; Drug: B
- B (Experimental): 14C GSK962040 (100 μg, SD, iv)
  Interventions: Drug: A

INTERVENTIONS:
Drug: A — GSK962040 (50 mg, SD, oral)
Drug: B — 14C GSK962040 (100 μg, SD, iv)
  Arms: A

SUMMARY:
The purpose of this study is to determine the absolute oral bioavailability and intravenous pharmacokinetics of GSK962040. The oral dose of 50 mg has been selected because it was well tolerated following single oral administration and it is considered to be within therapeutic dose range. The need to characterize the intravenous disposition of GSK962040 is in anticipation of drug use in special populations such as critically.

DETAILED DESCRIPTION:
GSK962040 is a selective non-peptide motilin receptor agonist which is being developed for the treatment of conditions associated with slow rates of gastric emptying. The purpose of this study is to determine the absolute bioavailability and the metabolic profile of GSK962040. Subjects will be administered a single oral dose of 50 mg followed by a single intravenous dose of 10 mL containing 100 microgram (not more than 270 nCi, 10 kBq) 14C GSK962040, administered by infusion over 15 minutes, beginning at 90 min after administration of the oral dose (approximate Cmax). The oral dose of 50 mg was well tolerated following single oral administration and is predicted to be a therapeutic dose. There is need to characterize GSK962040 disposition in anticipation of drug use in special populations such as critically ill patients. The intravenous (infused) microdose (100 microgram) is 500-fold lower than the oral dose, therefore exposure to GSK962040 originating from the infused microdose is considered negligible.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. In any case, liver function tests must be strictly within the normal range at screening.
* Male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Subjects must agree to use one of the contraception methods listed in Section 10.1. This criterion must be followed from the time of the first dose of study medication through at least 90 days following the dose of GSK962040.
* Body weight > or = 50 kg and BMI within the range 18.5-29.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec or QTc<480msec in subjects with Bundle Branch Block based on single or average QTc value of triplicate values obtained over a brief recording period.
* Normal physical examination (physical exam demonstrates no evidence of clinically active disease or physical or mental impairment). A subject with a clinical abnormality may be included only if the Principal Investigator or physician designee considers that the abnormality will not introduce additional risk factors and will not interfere with the study procedures. Consultation with the GSK medical monitor is required before such subjects may be included.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* .Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 3 months.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Consumption of red wine, Seville oranges, red wine, grapefruit or grapefruit juice, apple juice, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard), and charbroiled meats from 7 days prior to the dose of study medication. .
* Radiation exposure from clinical trials, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last twelve months or 10 mSv in the last five years.
* Subject has abnormal or altered upper gastrointestinal and/or biliary anatomy.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-06-14 (Actual); Primary Completion 2010-09-01 (Actual); Study Completion 2010-09-01 (Actual)

PRIMARY OUTCOMES:
PK parameters for GSK962040 following i.v. dose: AUC(0-inf), Cmax, tmax, t½, systemic clearance (CL), renal clearance (CLr), metabolic clearance (CLm), volume of distribution (Vss), and mean residence time (MRT). | 14 days
PK parameters following oral dose: AUC(0-inf), AUC(0-t), Cmax, tmax, t½, tlag, CLoral and absolute bioavailability (F). | 14 days

SECONDARY OUTCOMES:
Adverse Events | 14 days
Urine and fecal recovery of GSK962040 following a single oral and i.v. dose of [14C] GSK962040. | 14 days
Urine, fecal recovery and total recovery of radiocarbon (as a percentage of total radioactive dose in each interval and cumulative) | 14 days
Characterization and semi-quantitation of GSK962040-related metabolites in plasma, urine, and fecal homogenates following a single oral and i.v. dose of [14C] GSK962040. | 14 days
Vital signs | 14 days
ECGs | 14 days
Clinical lab assessments | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 114136 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114136?search=study&study_ids=114136#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register